CLINICAL TRIAL: NCT03533114
Title: A Double-blind, Placebo-controlled, Randomized Withdrawal, Multicenter Study of the Efficacy and Safety of JZP-258 in the Treatment of Idiopathic Hypersomnia (IH) With an Open-label Safety Extension
Brief Title: A Multicenter Study of the Efficacy and Safety of JZP-258 in the Treatment of Idiopathic Hypersomnia (IH) With an Open-label Safety Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JZP080-301; 2018-001311-79 (EudraCT Number)
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Idiopathic Hypersomnia
MeSH Terms: conditions — Idiopathic Hypersomnia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JZP-258 (Experimental): JZP-258 at the stable dose and regimen for 2 weeks.
  Interventions: Drug: JZP-258
- Placebo (Placebo Comparator): Placebo will be administered at a volume and regimen equivalent to the JZP-258 dose and regimen for 2 weeks.
  Interventions: Drug: Placebo Oral Solution

INTERVENTIONS:
Drug: JZP-258 — Participants randomized to JZP-258 will receive the dose taken at the end of the Stable Dose Period.
  Arms: JZP-258
Drug: Placebo Oral Solution — Participants randomized to Placebo will receive an oral solution at a volume and regimen equivalent to the JZP-258 dose taken at the end of the Stable Dose Period.
  Arms: Placebo

SUMMARY:
This is a study of the efficacy and safety of JZP-258, an oxybate mixed-salts oral solution being developed as a low sodium alternative product for Xyrem.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 75 years of age, inclusive, at the time of consent.
2. Have a primary diagnosis of IH according to the International Classification of Sleep Disorders ICSD-2 or ICSD-3 criteria.
3. At the Screening Visit and the Baseline Visit, subjects who are not on Xyrem at study entry must have ESS scores ≥ 11 (as assessed with a look-back period of 1 week).
4. If currently treated with Xyrem, must have documented clinical improvement of EDS after the initiation of Xyrem per Investigator's clinical judgment.
5. Average nightly total sleep time of ≥ 7 hours, per subject history. Average nightly total sleep time will be confirmed by Investigator's review of sleep diaries collected during the final 2 weeks of the Screening Period.
6. If currently treated with stimulants and / or alerting agents or nicotine replacement therapy, must have been taking the same regimen and dose for at least 2 months prior to screening and must agree to take the same dose leading up to and throughout the Double-blind Randomized Withdrawal Period.
7. Have used a medically acceptable method of contraception for at least 2 months prior to the first dose of study drug and consent to use a medically acceptable method of contraception from the first dose of study drug, throughout the entire study period, and for 90 days after the last dose of study drug.

Exclusion Criteria:

1. Hypersomnia due to another medical, behavioral, or psychiatric disorder condition.
2. Evidence of untreated or inadequately treated sleep-disordered breathing.
3. Clinically significant parasomnias (eg, sleep walking, rapid eye movement sleep behavior disorder, etc.).
4. Current or past (within 1 year) major depressive episode according to DSM-5 criteria. Patients with depression under control are allowed per the judgment of the Investigator or the treating physician and the anti-depressant treatment has to be stable for at least 6 months prior to Screening and remain stable for the duration of the study.
5. Current suicidal risk as determined from history by presence of active suicidal ideation as indicated by positive response to item #4 or #5 on C-SSRS, or any history of suicide attempt.
6. Occupation requiring nighttime shift work or variable shift work with early work start times or other occupations that could affect the safety of the subject per the judgment of the Investigator.
7. Treatment or planned treatment with any CNS sedating agents, including but not limited to benzodiazepines or other sedating anxiolytics, sedating antidepressants, hypnotics, sedatives, neuroleptics, opoids, barbiturates, phenytoin, melatonin, ethosuximide, medications containing valproic acid or its sodium salt, or any other medication in which the subject experiences sedation are prohibited during the study. Treatment must have been discontinued within 2 weeks or 5 half-lives, whichever is longer, prior to enrollment. The Investigator must ensure that discontinuation from these medications is medically supervised. Subjects must abstain from these medications during the study.
8. Current or past substance use disorder (including alcohol) according to DSM-5 criteria, or the subject is unwilling to refrain from consuming alcohol, cannabinoids, or prohibited medications during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (40):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Wright Clinical Research, LLC, Birmingham, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Mayo Clinic Building, Phoenix, Arizona
  - Southern California Institute for Respiratory Diseases, Inc., Los Angeles, California
  - Stanford Sleep Medicine Center, Redwood City, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Delta Waves, Inc., Colorado Springs, Colorado
  - PAB Clinical Research, Brandon, Florida
  - Suncoast Research Group, Miami, Florida
  - Bio-Medical Research, LLC, Miami, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - NeuroTrials Research, Atlanta, Georgia
  - Sleep Practitioners, LLC, Macon, Georgia
  - SleepCare Research Institute d/b/a Clinical Research, Stockbridge, Georgia
  - Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Baystate Wesson Sleep Clinic, Springfield, Massachusetts
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Clinical Neurophysiology Services, P.C., Sterling Heights, Michigan
  - Minnesota Lung Center, Minneapolis, Minnesota
  - Clayton Sleep Institute, LLC, St Louis, Missouri
  - Montefiore Medical Center/Sleep-Wake Disorders Center, The Bronx, New York
  - American Health Research, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Research Carolina, Huntersville, North Carolina
  - Clinical Research of Lake Norman, Mooresville, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Intrepid Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Sleep Medicine and Neuroscience Institute, Dublin, Ohio
  - Lynne Health Science Institute, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - Neurology Clinic, PC, Cordova, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
- Belgium (3):
  - Anima Research Center, Alken
  - Antwerp University Hospital, Edegem
  - CHU UCL Namur site de Sainte Elisabeth, Namur
- Czechia (3):
  - Nemocnice Ceske Budejovice a.s., České Budějovice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
- VitalMed Oy, Helsinki, Finland
- France (5):
  - CHU de Grenoble - Hôpital Michallon, Grenoble
  - Hopital Roger Salengro, Lille
  - Hopital Gui de Chauliac, Montpellier
  - CHU Nantes - Hopital Nord Laënnec, Nantes
  - Hopital Pitie-Salpetriere, Paris
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Osrodek Badan Klinicznych CROMED, Poznan
  - lnstytut Psychiatrii i Neurologii, Zaklad Neurofizjologii Klinicznej, Warsaw
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Vithas Nuestra Señora de America, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Araba, Vitoria-Gasteiz
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bogan RK, Fuller DS, Whalen M, Casstevens C, Schneider LD. A minimal clinically important difference for the sleep inertia visual analog scale in idiopathic hypersomnia. J Clin Sleep Med. 2025 Jul 1;21(7):1209-1216. doi: 10.5664/jcsm.11662. PMID 40135693
- [Derived] Morse AM, Dauvilliers Y, Arnulf I, Thorpy MJ, Foldvary-Schaefer N, Chandler P, Chen A, Hickey L, Black J, Bogan RK. Long-term efficacy and safety of low-sodium oxybate in an open-label extension period of a placebo-controlled, double-blind, randomized withdrawal study in adults with idiopathic hypersomnia. J Clin Sleep Med. 2023 Oct 1;19(10):1811-1822. doi: 10.5664/jcsm.10698. PMID 37409509
- [Derived] Dauvilliers Y, Arnulf I, Foldvary-Schaefer N, Morse AM, Sonka K, Thorpy MJ, Mignot E, Chandler P, Parvataneni R, Black J, Sterkel A, Chen D, Skobieranda F, Bogan RK. Safety and efficacy of lower-sodium oxybate in adults with idiopathic hypersomnia: a phase 3, placebo-controlled, double-blind, randomised withdrawal study. Lancet Neurol. 2022 Jan;21(1):53-65. doi: 10.1016/S1474-4422(21)00368-9. PMID 34942138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The safety population is categorized according to the presence or absence of medications used to treat IH symptoms at the time of study baseline.
Groups:
- On Baseline IH Medication: Participants treated with medication for IH at baseline.
- Treatment Naive: Participants not treated with medication for IH at baseline.
Period: Overall
Arm/Group | On Baseline IH Medication | Treatment Naive
Started | 88 | 66
Completed | 57 | 38
Not Completed | 31 | 28
Not completed — Adverse Event | 16 | 11
Not completed — Consent Withdrawal by Participant | 7 | 6
Not completed — Lack of Efficacy | 5 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Protocol deviation | 1 | 1
Not completed — Failure to meet randomization criteria | 1 | 2
Not completed — Non-Compliance with study drug | 0 | 1
Not completed — Other | 0 | 1
Period: Open Label Titration and Optimization
Arm/Group | On Baseline IH Medication | Treatment Naive
Started | 88 | 66
Completed | 72 | 53
Not Completed | 16 | 13
Not completed — Adverse Event | 11 | 8
Not completed — Consent Withdrawal by Participant | 2 | 1
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Deviation | 0 | 1
Not completed — Non-Compliance with Study Drug | 0 | 1
Period: Stable Dose
Arm/Group | On Baseline IH Medication | Treatment Naive
Started | 71 | 52
Completed | 69 | 50
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Consent Withdrawal by Participant | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Period: Double Blind Randomized-Withdrawal
Arm/Group | On Baseline IH Medication | Treatment Naive
Started | 69 | 47
JZP-258 | 57 | 0
Placebo | 0 | 59
Completed | 67 | 46
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Failure to Meet Randomization Criteria | 1 | 0
Period: Open-Label Safety Extension
Arm/Group | On Baseline IH Medication | Treatment Naive
Started | 65 | 41
Completed | 57 | 38
Not Completed | 8 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Consent Withdrawal by Participant | 2 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Naïve: Participants not treated with medication for IH at baseline.
- Total: Total of all reporting groups
Arm/Group | On Baseline IH Medication | Treatment Naïve | Total
Number analyzed (Participants) | 88 | 66 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (13.37) | 39.4 (14.25) | 40.3 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 40 | 105
  Male | 23 | 26 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 4 | 9
  White | 76 | 53 | 129
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  North America | 69 | 35 | 104
  Europe | 19 | 31 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Epworth Sleepiness Scale (ESS) Score
Description: The ESS is a 8-item self reported questionnaire intended to measure daytime sleepiness. In this test, participants answer questions with regard to the level of sleepiness they experienced over approximately the 7 days prior to the assessment while performing eight common, non-stimulating activities. The ESS total score range is 1 to 24. Each activity is rated on a 4-point scale ranging from a minimum of "would never doze" to a maximum of "a high chance of dozing." Thus, the ESS scale range is as follows: 0=would never doze, 1=slight chance of dozing, 2=moderate chance of dozing, 3=high chance of dozing; 0 indicates a better outcome, and 3 indicates a worse outcome. A positive mean change value indicates an increase in score from the end of the stable dose period and worsened daytime sleepiness. A higher ESS score (above 10) reflects a greater average sleep propensity in daily life (ASP) , or daytime sleepiness.
Time Frame: Change from the end of the Stable Dose Period to the end of the Double-blind Randomized Withdrawal Period (DBRW) (2 Weeks)
Population: The Modified Intent to Treat (mITT) analysis set included all participants who were randomized to JZP258 or placebo, who received at least 1 dose of study drug during the DBRW and have had at least one set of post randomization assessments for ESS or IHSS, or a PGIc value at the end of the DBRW.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- JZP-258: Participants randomized to JZP-258 will receive the dosing regimen taken during the Stable Dose Period.
- Placebo: Participants randomized to placebo will receive an oral solution equivalent to the dosing regimen of JZP-258 taken during the Stable Dose Period.
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 56 | 59
score on a scale | 0.7 (3.22) | 7.4 (5.16)

2. Secondary Outcome: Percentage of Participants Reported as Worse on the Patient Global Impression of Change (PGIc)
Description: The Patient Global Impression - Change (PGIc) scale was completed by the participant. The PGI-C scale rated the participant's condition at a specified time point on a 7-point scale ranging from a minimum of "Very much improved" to a maximum of "Very much worse." The PGIc scale consists of the following ratings: 1-Very Much improved, 2-Much improved, 3-Minimally improved, 4-No change, 5-Minimally worse, 6-Much worse, 7-Very much worse; a rating of 1 indicates a better outcome, and a rating of 7 indicates a worse outcome. Worsened condition was defined as a PGIc rating of 5, 6, or 7.
Time Frame: At the end of the DBRW Period (2 Weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 56 | 59
participants | 12 | 52

3. Secondary Outcome: Change in Total Score on the Idiopathic Hypersomnia Severity Scale (IHSS)
Description: The IHSS is a 14-item self-reported questionnaire assessing the severity of IH symptoms of excessive sleepiness, prolonged sleep duration, cognitive impairment and sleep inertia. Total scores can range from 0 to 50, with higher scores indicating a greater severity or frequency of symptoms.
Time Frame: Change from the end of the Stable Dose Period to the end of the DBRW Period (2 Weeks)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 56 | 59
score on a scale | 0.0 [-8 to 24] | 14.0 [-2 to 38]

4. Secondary Outcome: Percentage of Participants Reported as Worse on the Clinical Global Impression of Change (CGIc)
Description: The CGIc scale is a 7-point Likert-type scale that rates the Investigator's impression of any change in the severity of the participant's condition at a specified time point. The participant was rated on a 7-point scale ranging from a minimum of "Very much improved" to a maximum of "Very much worse." The CGIc scale consists of the following ratings: 1-Very Much improved, 2-Much improved, 3-Minimally improved, 4-No change, 5-Minimally worse, 6-Much worse, 7-Very much worse; a rating of 1 indicates a better outcome, and a rating of 7 indicates a worse outcome. Worsened condition was defined as a CGIc rating of 5, 6, or 7.
Time Frame: At the end of the DBRW Period (2 Weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 56 | 59
participants | 12 | 52

5. Secondary Outcome: Change in Total Score on the Functional Outcomes of Sleep Questionnaire (FOSQ-10)
Description: The FOSQ-10 is a short version of the original FOSQ-30 instrument, which is a disease specific quality of life questionnaire to determine functional status in adults. Measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these activities are improved by effective treatment. The questionnaire has a 4-point Likert response format (e.g., 1= extreme difficulty, 2= moderate difficulty, 3=a little difficulty, and 4 =no difficulty). FOSQ-10 total score is calculated by first taking the mean of the items for each subscale with more than 1 item completed and then taking the mean across the non-missing 5 subscales (General Productivity, Activity Level, Vigilance, Social Outcomes, Intimacy and Sexual Relationship) multiplied by 5. The score ranges from a minimum of 5 points to a maximum of 20 points, with higher scores indicating better functional status.
Time Frame: Change from the end of the Stable Dose Period to the end of the DBRW Period (2 Weeks)
Population: The Modified Intent to Treat (mITT) analysis set included all participants who were randomized to JZP258 or placebo, who received at least 1 dose of study drug during the DBRW and have had at least one set of post randomization assessments for ESS or IHSS, or a PGIc value at the end of the DBRW. JZP-258 overall number was 54 and placebo group overall number was 56 as fewer participants were available for this particular assessment.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 54 | 56
score on a scale | -0.08 [-8.5 to 4.5] | -4.17 [-12.5 to 1.3]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were recorded from the time on or after the first dose of study drug, including adverse events that occurred until 30 days after the last dose date up to 42 weeks.
Groups:
- JZP-058: Participants randomized to JZP-258 will receive the dose taken at the end of the Stable Dose Period at the stable dose and regimen for 2 weeks.
- Placebo: Participants randomized to placebo were administered placebo oral solution at a volume and regimen equivalent to the JZP-258 dose and regimen for 2 weeks.
Arm/Group | On Baseline IH Medication | Treatment Naive | JZP-058 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/66 | 0/154 | 0/59
Serious Adverse Events (participants affected / at risk) | 2/88 | 2/66 | 4/154 | 0/59
Other Adverse Events (participants affected / at risk) | 64/88 | 39/66 | 97/154 | 10/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Baseline IH Medication (N=88) | Treatment Naive (N=66) | JZP-058 (N=154) | Placebo (N=59)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (5) | 1 (5) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Baseline IH Medication (N=88) | Treatment Naive (N=66) | JZP-058 (N=154) | Placebo (N=59)
Diarrhoea (Gastrointestinal disorders) | 11 (15) | 3 (4) | 12 (17) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 2 (2) | 10 (10) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (31) | 13 (14) | 34 (44) | 1 (1)
Vomiting (Gastrointestinal disorders) | 15 (18) | 3 (3) | 17 (19) | 2 (2)
Fatigue (General disorders) | 8 (10) | 4 (5) | 11 (14) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (7) | 12 (13) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 5 (6) | 12 (13) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (7) | 6 (7) | 12 (14) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 7 (7) | 14 (14) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (9) | 1 (1) | 8 (10) | 0 (0)
Dizziness (Nervous system disorders) | 8 (8) | 11 (11) | 19 (19) | 0 (0)
Headache (Nervous system disorders) | 15 (26) | 12 (16) | 27 (40) | 2 (2)
Tremor (Nervous system disorders) | 9 (11) | 0 (0) | 9 (11) | 0 (0)
Anxiety (Psychiatric disorders) | 10 (11) | 8 (8) | 17 (18) | 1 (1)
Insomnia (Psychiatric disorders) | 13 (15) | 4 (4) | 11 (13) | 6 (6)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (10) | 2 (2) | 9 (12) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 5 (6) | 4 (5) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT03533114/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT03533114/SAP_001.pdf